CLINICAL TRIAL: NCT02276664
Title: Capitalizing on a Teachable Moment to Promote Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: MCC-17952; 4KB05 (Other: James and Esther King Biomedical Research Program)
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Smoking Cessation
Keywords: lung cancer prevention
MeSH Terms: conditions — Smoking Cessation | interventions — National Health Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study 1 - Focus Groups (No Intervention): Using focus group methodology, investigators will identify and explore new content topics for inclusion in smoking cessation booklets and gather feedback about the existing Stop Smoking for Good booklets regarding tone and message design. Results will be used to modify and adapt the existing cessation intervention.
- Study 2 - Self-Help Intervention (SHI) (Experimental): The SHI arm will receive the intervention developed in Study I.
  Interventions: Behavioral: Self-Help (SHI)
- Study 2 - Usual Care (UC) (Active Comparator): The UC arm will receive the existing Clearing the Air smoking-cessation manual.
  Interventions: Behavioral: Usual Care (UC)

INTERVENTIONS:
Behavioral: Self-Help (SHI) — The newly revised Stop Smoking for Good booklets.
  Arms: Study 2 - Self-Help Intervention (SHI)
Behavioral: Usual Care (UC) — The existing Clearing the Air smoking-cessation manual published by the National Cancer Institute (NCI).
  Arms: Study 2 - Usual Care (UC)

SUMMARY:
The purpose of this study is to develop and test a self-help smoking cessation treatment for patients receiving a lung cancer screening computed tomography (CT) scan.

DETAILED DESCRIPTION:
Conduct Formative Research (Months 1 - 4): Identification of emergent themes and responses to existing booklets.

Adapt and Refine Booklets (Months 5 - 8): Advanced drafts of booklets.

Final Reactions to Draft Booklets (Months 9 - 12): Series of smoking cessation booklets for spiral computed tomography (CT) patients.

ELIGIBILITY:
Inclusion Criteria:

Study 1

* Participants for Study I will be drawn from a list of patients who have received a CT scan at the Moffitt Cancer Center
* Smoked at least one cigarette per week prior to undergoing the CT scan
* Able to speak and read English

Study 2

* Smoked at least one cigarette over the past week
* Able to read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Study 1 - Completion of Formative Evaluation | Up to 12 months
  Complete formative research to adapt and refine the existing Stop Smoking for Good booklets.
Study 2 - Rate of Seven-Day Abstinence | Seven-day abstinence will be assessed at each follow-up, allowing for calculation of point-prevalence abstinence rates. For this pilot, we will not bioverify self-reported abstinence.
  Up to 9 months

SECONDARY OUTCOMES:
Rate of Intervention Demand | Up to 9 months
  Demand will be estimated by noting accrual rates into the study.
Degree of Practicality | Up to 9 months
  Practicality encompasses the degree to which investigators are able to carry out all the piloted elements of the planned randomized control trial (RCT) successfully and efficiently (i.e., recruitment, screening, randomization, and follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Brandon, Ph.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H Lee Moffitt Cancer Center, Tampa, Florida, United States